CLINICAL TRIAL: NCT07034898
Title: A Randomized Comparative Study of Dexmedetomidine Versus Labetalol in Attenuating Airway Stress Response in Hypertensive Patients Undergoing Craniotomy
Brief Title: Dexmedetomidine vs Labetalol for Airway Stress in Hypertensive Craniotomy Patients
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MS /806/2024
Record Dates: First submitted 2025-06-15; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-02

CONDITIONS: Airway Stress Response
Keywords: Airway Stress Response; Extubation; Dexmedetomidine; Labetalol; Hemodynamic Stability; Hypertension; Craniotomy
MeSH Terms: conditions — Hypertension | interventions — Dexmedetomidine; Adrenergic alpha-2 Receptor Agonists; Labetalol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine Group (Experimental): A 50 mL syringe pump containing 0.5 mcg/kg dexmedetomidine diluted with saline to 50 mL will be infused at 300 mL/hr to complete within 10 minutes, followed by extubation.
  Interventions: Drug: Dexmedetomidine
- Labetalol Group (Experimental): A 50 mL syringe pump containing 0.5 mg/kg labetalol diluted with saline to 50 mL will be infused at 300 mL/hr to complete within 10 minutes, followed by extubation.
  Interventions: Drug: Labetalol

INTERVENTIONS:
Drug: Dexmedetomidine — Participants in this arm will receive dexmedetomidine at a dose of 0.5 mcg/kg, diluted with normal saline to a total volume of 50 mL. The solution will be administered intravenously via a syringe pump at an infusion rate of 300 mL/hour, completing over 10 minutes immediately prior to extubation.
  Other Names: Precedex; DEX; Alpha-2 agonist
  Arms: Dexmedetomidine Group
Drug: Labetalol — Participants in this arm will receive labetalol at a dose of 0.5 mg/kg, diluted with normal saline to a total volume of 50 mL. The solution will be administered intravenously via a syringe pump at an infusion rate of 300 mL/hour, completing over 10 minutes immediately prior to extubation.
  Other Names: Normodyne; Trandate; LAB; Alpha/Beta blocker
  Arms: Labetalol Group

SUMMARY:
This randomized trial compares dexmedetomidine and labetalol in controlling airway and hemodynamic stress during extubation in hypertensive patients undergoing craniotomy. Outcomes include extubation quality, vital signs, sedation, and adverse effects.

DETAILED DESCRIPTION:
A. Preoperative Settings:

Patients will undergo standard pre-anesthetic assessment, including review of medical history, fasting status, and laboratory investigations. Eligibility will be confirmed based on inclusion and exclusion criteria. After obtaining informed consent, patients will be randomly assigned into two groups using a computer-generated randomization table and sealed envelopes.

B. Intraoperative and Postoperative Settings:

All patients will receive standardized general anesthesia with continuous monitoring. Following completion of surgery and while still under anesthesia, the study drug (either dexmedetomidine or labetalol) will be administered over 10 minutes. Extubation will be performed thereafter.

Hemodynamic parameters including arterial blood pressure and heart rate will be recorded at baseline, during drug administration, and at specific intervals post-extubation. Extubation quality will be assessed using a five-point scale, and sedation levels using the Richmond Agitation-Sedation Scale. Adverse events such as hypotension, bradycardia, or respiratory issues will be documented and managed as per protocol.

This structured approach aims to evaluate which agent provides better control of stress responses during emergence from anesthesia in hypertensive patients undergoing craniotomy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30 and 60 years

American Society of Anesthesiologists (ASA) physical status II

Diagnosed hypertension

Scheduled for elective craniotomy under general anesthesia

Able and willing to provide informed consent

Exclusion Criteria:

* ASA physical status III or IV

Uncontrolled comorbidities (e.g., diabetes mellitus)

Coagulopathy or current use of anticoagulant or antiplatelet therapy

Known allergy or hypersensitivity to dexmedetomidine or labetalol

Emergency craniotomy

Pregnant or breastfeeding women

Patients with a history of severe cardiac arrhythmias

Inability to provide informed consent

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Extubation Assessed Using a Standardized 5-Point Scale | Within the first 5 minutes after extubation
  Extubation quality will be assessed immediately after extubation using a standardized 5-point scale, where:
  1. = No cough, smooth extubation
  2. = Minimal coughing (1-2 times), smooth extubation
  3. = Moderate coughing (3-4 times)
  4. = Severe coughing (5-10 times) or difficulty breathing
  5. = Poor extubation, very uncomfortable, forced breathing (e.g., laryngospasm or coughing >10 times)
  A lower score indicates better extubation quality. The outcome will be evaluated by a blinded observer within the first 5 minutes post-extubation.

SECONDARY OUTCOMES:
Sedation Level Post-Extubation | Within 10 minutes after extubation
  Sedation level will be evaluated using the Richmond Agitation-Sedation Scale (RASS) within 10 minutes following extubation. The RASS is a validated tool for assessing the level of consciousness in patients, with scores ranging from +4 (combative) to -5 (unarousable). A score of 0 indicates an alert and calm state, while negative scores represent increasing levels of sedation and positive scores reflect agitation.
Mean Arterial Pressure (MAP) Variation from Baseline | From baseline (pre-infusion) to 5 minutes post-extubation
  Mean Arterial Pressure (MAP) will be recorded at baseline (pre-drug administration), during drug infusion, immediately post-extubation, and at 1, 3, and 5 minutes after extubation. The goal is to evaluate the extent to which MAP deviates from baseline values following administration of either dexmedetomidine or labetalol. MAP stability is defined as values maintained within ±20% of baseline. This outcome will be used to assess the effectiveness of each drug in attenuating hemodynamic responses associated with extubation in hypertensive patients undergoing craniotomy.
Heart Rate Variation from Baseline | From baseline (pre-infusion) to 5 minutes post-extubation.
  Heart rate (HR) will be recorded at baseline (prior to administration of the study drug), during drug infusion, immediately after extubation, and at 1, 3, and 5 minutes post-extubation. The primary objective is to compare heart rate responses between the dexmedetomidine and labetalol groups and determine how effectively each drug maintains HR within ±20% of the baseline. This outcome will help evaluate the efficacy of both interventions in attenuating the sympathetic response to extubation in hypertensive patients undergoing craniotomy.
Incidence of Adverse Events During and After Extubation | From initiation of drug infusion to 10 minutes post-extubation
  Adverse events will be monitored and documented from the start of study drug administration until 10 minutes post-extubation. Events of interest include bradycardia (heart rate < 50 bpm), hypotension (MAP decrease > 20% from baseline), respiratory depression, laryngospasm, severe coughing, nausea, vomiting, or any other clinically significant complication. All adverse events will be recorded, classified by severity, and managed according to standard anesthetic protocols. This outcome aims to compare the safety profiles of dexmedetomidine and labetalol in the context of emergence from anesthesia in hypertensive patients undergoing craniotomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared once study is completed
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Before 3/2026
Access Criteria: Free